CLINICAL TRIAL: NCT03792425
Title: Clinical Evaluation of Pink Esthetic Score Following Delayed Implant Placement With Connective Tissue Graft With and Without Temporization in the Maxillary Esthetic Zone With Thin Gingival Biotype
Brief Title: Clinical Evaluation of Pink Esthetic Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha fawzy el sayed ali abd allah, Teaching assistant at el Ahram canadian university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2121992
Record Dates: First submitted 2018-12-27; First posted 2019-01-03 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Thin Gingiva

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implant with immediate temporization (Other): Immediate nonfunctional loading
  Interventions: Procedure: Connective tissue graft and implant placement
- Delayed implant without temporization (Other): Conventional loading protocol
  Interventions: Procedure: Connective tissue graft and implant placement

INTERVENTIONS:
Procedure: Connective tissue graft and implant placement — Augmenting soft tissue with connective tissue graft

SUMMARY:
Clinical evaluation of pink esthetic score in delayed implants in thin gingival biotype with and without temporization in the esthetic zone

DETAILED DESCRIPTION:
Clinical evaluation of the pink esthetic score with and withiut temporization in thin gingival biotype in the maxillary esthetic zone with subepithelial connective tissue graft in bith groups

ELIGIBILITY:
Inclusion Criteria:

* patients with missing teeth in the maxillary esthetic zone with thin gingival biotype and adequate arch space

Exclusion Criteria:

* deficient ridge , crowns on the adjacent teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Pink esthetic score | 1 year from the base line
  Clinical assessment accotding to furhausser et al

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Fawzy M, Hosny M, El-Nahass H. Evaluation of esthetic outcome of delayed implants with de-epithelialized free gingival graft in thin gingival phenotype with or without immediate temporization: a randomized clinical trial. Int J Implant Dent. 2023 Feb 13;9(1):5. doi: 10.1186/s40729-023-00468-0. PMID 36781590